CLINICAL TRIAL: NCT00691938
Title: A Phase I/II Study of LBH589 Plus Decitabine for Patients Age ≥ 60 Years With High Risk MDS or AML
Brief Title: LBH589 Plus Decitabine for Myelodysplastic Syndromes (MDS) or Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0172 / 201012979
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: LBH589; Decitabine; panobinostat; histone deacetylase; methylation; hypomethylation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Panobinostat; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Level 1 (Experimental): LBH589 10 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  Interventions: Drug: LBH589; Drug: Decitabine
- Level 2 (Experimental): LBH589 15 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  Interventions: Drug: LBH589; Drug: Decitabine
- Level 3 (Experimental): LBH589 20 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  Interventions: Drug: LBH589; Drug: Decitabine
- Level 4 (Experimental): LBH589 30 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  Interventions: Drug: LBH589; Drug: Decitabine
- Level 5 (Experimental): LBH589 40 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  Interventions: Drug: LBH589; Drug: Decitabine
- Level 5B (Experimental): LBH589 40 mg/day three times a week on nonconsecutive days for the first 2 weeks in a 28 day cycle.
  Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  Interventions: Drug: LBH589; Drug: Decitabine
- Phase II (Experimental): LBH589 will be given in the dose and in the schedule that was found to work in the Phase I portion which was Level 5B.
  Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  Interventions: Drug: LBH589; Drug: Decitabine

INTERVENTIONS:
Drug: LBH589
  Other Names: Panobinostat
Drug: Decitabine
  Other Names: Dacogen; 5-aza-2'-deoxycytidine

SUMMARY:
This study is designed to evaluate the combination of LBH589 and decitabine in patients age ≥ 60 years with high risk Myelodysplastic Syndrome (IPSS Int-2 or High) or Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
To address the need for less toxic, more effective treatments for older patients with advanced MDS and AML, the purpose of this Phase 1-2 single institution study is to evaluate the safety and efficacy of LBH 589 and decitabine administered in combination.

Decitabine is an epigenetic modifier of gene expression that has been shown to be well-tolerated in this population at the dose schedule proposed in this study, with reasonable efficacy. Although its precise mechanism of action is incompletely understood, it is postulated to work by reactivating the expression of key tumor suppressor genes silenced in tumor cells by reversing a pattern of hypermethylation of promotor elements.

LBH389 is likewise an epigenetic modifier that inhibits the deacetylation of both histones and non-histone proteins, including HSP90 and p53. Although clinical experience with LBH589 in AML is limited, aberrant histone deacetylase activity has been previously shown to play a significant role in the pathogenesis of AML. The addition of LBH589 to a decitabine regimen of previously established efficacy and tolerability will allow us to evaluate the hypothesis that two epigenetic modifiers that are believed to work through distinct mechanisms of action may act together to improve the responses of patients treated with decitabine alone, without significant additional toxicity.

ELIGIBILITY:
Inclusion Criteria:

* AML (except t(15;17), inv(16) or t(8;21) and variants) or high risk MDS (IPSS Int-2 or High) diagnosed according to WHO criteria (see Appendix 1)
* Age ≥ 60 years old
* Not a candidate for allogeneic stem cell transplantation within next 12 weeks
* Ability to provide written informed consent, obtained prior to participation in the study and any related procedures being performed
* Patients must meet the following laboratory criteria:
* Serum albumin ≥ 3 g/dL
* Aspartate aminotransferase (AST)/SGOT and alanine aminotransferase (ALT)/SGPT ≤ 2.5 x upper limit of normal (ULN) ) or ≤ 5.0 x ULN if the transaminase elevation is due to leukemic involvement
* Serum bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
* Serum potassium ≥ lower limit of normal (LLN)
* Serum phosphorus ≥ LLN
* Serum total calcium (corrected for serum albumin) or serum ionized calcium ≥ LLN
* Serum magnesium ≥ LLN, thyroid stimulating hormone (TSH) and free thyroxine (T4) within normal limits (WNL) (patients may be on thyroid hormone replacement)
* Baseline MUGA or ECHO must demonstrate left ventricular ejection fraction (LVEF) ≥ the lower limit of the institutional normal.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2

Exclusion Criteria:

* Prior treatment for MDS / AML with Histone deacetylase (HDAC) inhibitor or hypomethylating agent (e.g., Decitabine, azacitidine etc.)
* Active central nervous system (CNS) involvement with MDS/AML
* Impaired cardiac function including any one of the following:
* Screening electrocardiogram (ECG) with a QTc > 450 msec confirmed by central laboratory prior to enrollment to the study
* Patients with congenital long QT syndrome
* History of sustained ventricular tachycardia
* Any history of ventricular fibrillation or torsades de pointes
* Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible.
* Patients with a myocardial infarction or unstable angina within 6 months of study entry
* Congestive heart failure (NY Heart Association class III or IV)
* Right bundle branch block and left anterior hemiblock (bifasicular block)
* Uncontrolled hypertension
* Concomitant use of drugs with a risk of causing torsades de pointes
* Patients with unresolved diarrhea > CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have received chemotherapy or any investigational drug < 2 weeks or hydroxyurea < 48 hours prior to starting study drug or who have not recovered from side effects of such therapy.
* Concomitant use of any anti-cancer therapy or radiation therapy
* Male patients whose sexual partners are women of child bearing potential (WOCBP) not using effective birth control
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
* Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-06; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Uy, M.D., Principal Investigator — Washington Univerisity
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Cashen, A., G. J. Schiller, et al. (2006). Phase II Study of Low-Dose Decitabine for the Front-Line Treatment of Older Patients with Acute Myeloid Leukemia (AML). ASH Annual Meeting Abstracts 108(11): 1984.
- [Derived] Uy GL, Duncavage EJ, Chang GS, Jacoby MA, Miller CA, Shao J, Heath S, Elliott K, Reineck T, Fulton RS, Fronick CC, O'Laughlin M, Ganel L, Abboud CN, Cashen AF, DiPersio JF, Wilson RK, Link DC, Welch JS, Ley TJ, Graubert TA, Westervelt P, Walter MJ. Dynamic changes in the clonal structure of MDS and AML in response to epigenetic therapy. Leukemia. 2017 Apr;31(4):872-881. doi: 10.1038/leu.2016.282. Epub 2016 Oct 14. PMID 27740633
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 06/23/2008 and closed to participant enrollment on 11/06/2012.
Groups:
- Level 1: LBH589 10 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m2 IV on days 1-5 in a 28 day cycle.
- Level 2: LBH589 15 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m2 IV on days 1-5 in a 28 day cycle.
- Level 3: LBH589 20 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m2 IV on days 1-5 in a 28 day cycle.
- Level 4: LBH589 30 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m2 IV on days 1-5 in a 28 day cycle.
- Level 5: LBH589 40 mg/day three times a week on nonconsecutive days in a 28 day cycle.
  Decitabine 20 mg/m2 IV on days 1-5 in a 28 day cycle.
- Level 5B: LBH589 40 mg/day three times a week on nonconsecutive days for the first 2 weeks in a 28 day cycle.
  Decitabine 20 mg/m2 IV on days 1-5 in a 28 day cycle.
- Phase II: LBH589 will be given in the dose and in the schedule that was found to work in the Phase I portion which was dose from Level 5B.
  Decitabine 20 mg/m2 IV on days 1-5 in a 28 day cycle.
Period: Overall Study
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4 | Level 5 | Level 5B | Phase II
Started | 5 | 3 | 6 | 8 | 10 | 6 | 14
Completed | 4 | 3 | 6 | 8 | 10 | 6 | 14
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — QTc prolongation | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4 | Level 5 | Level 5B | Phase II | Total
Number analyzed (Participants) | 5 | 3 | 6 | 8 | 10 | 6 | 14 | 52
Age, Continuous [Median (Full Range); unit: years] | 69 [62 to 74] | 69 [67 to 83] | 68 [62 to 75] | 72 [61 to 86] | 73 [64 to 87] | 71 [63 to 80] | 66 [61 to 78] | 70 [61 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 3 | 2 | 5 | 10 | 27
  Male | 2 | 2 | 3 | 5 | 8 | 1 | 4 | 25
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 6 | 8 | 10 | 6 | 14 | 52

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of LBH589 When Given in Combination With Decitabine
Time Frame: Completion of Phase I enrollment for MTD (approximately 26 months)
Population: After enrolling all Phase I patients in Dose Levels 1-5b, the maximum tolerated dose was not determined. The Phase II portion of the study used the 5b dose level.
Measure: Number; unit: mg (level 5b dosing schedule)
Arm/Group | Phase I (Includes Levels 1-5)
Number analyzed (Participants) | 37
mg (level 5b dosing schedule) | 40

2. Primary Outcome: Phase II: Overall Rate of Morphologic Complete Remission (CR) + Cytogenetic Complete Remission (CRc) + Morphologic Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: * Morphologic complete remission (CR). A CR designation requires that the patient achieve the morphologic leukemia-free state with less than 5% blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. There should be no blasts with Auer rods or persistence of extramedullary disease. Patients must also have an absolute neutrophil count of more than 1,000/μLand platelets of 100,000/μL.
  * Cytogenetic complete remission (CRc). A CRc will be defined by the achievement of a CR with reversion to a normal karyotype in a minimum of 20 metaphases analyzed by cytogenetics.
  * Morphologic complete remission with incomplete blood count recovery (CRi): Achievement of all of the criteria for CR except for residual neutropenia (< 1,000/μL) or thrombocytopenia (< 100,000/μL).
Time Frame: Up to 12 months
Measure: Number; unit: percentage of participants
Groups:
- Level 1-Phase II (All Patients Enrolled): * Level 1:LBH589 10 mg/day three times a week on nonconsecutive days in a 28 day cycle. Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  * Level 2:LBH589 15 mg/day three times a week on nonconsecutive days in a 28 day cycle. Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  * Level 3: LBH589 20 mg/day three times a week on nonconsecutive days in a 28 day cycle. Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  * Level 4:LBH589 30 mg/day three times a week on nonconsecutive days in a 28 day cycle. Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  * Level 5:LBH589 40 mg/day three times a week on nonconsecutive days in a 28 day cycle. Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
  * Level 5B/Phase II:LBH589 will be given in the dose and in the schedule that was found to work in the Phase I portion which was dose from Level 5B. Decitabine 20 mg/m^2 IV on days 1-5 in a 28 day cycle.
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 51
percentage of participants | 11.8

3. Secondary Outcome: Rate of Cytogenetic Complete Remission (CRc)
Description: Cytogenetic complete remission (CRc). A CRc will be defined by the achievement of a CR with reversion to a normal karyotype in a minimum of 20 metaphases analyzed by cytogenetics.
Time Frame: Up to 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 51
percentage of participants | 3.9

4. Secondary Outcome: Changes in Quality of Life Scores as Measured by the Function Assessment of Cancer Therapy-Leukemia (FACT-Leu) Version 4
Description: -The FACT-Leu consists of a 27-item compilation of general questions divided into four primary quality of life domains: physical well-being, social/family well being, emotional well-being, and functional well-being along with a 17 item subscale developed specifically for patients with leukemia.
Time Frame: Up to approximately 12 months after start of treatment
Population: Data was not collected for this outcome measure.
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Response
Description: Time to response is defined as the date of the first dose of study drug to the date that all criteria for CR or CRi are fulfilled.
Time Frame: Up to 12 months
Population: Number of participants analyzed are participants that met the criteria for CR or CRi.
Measure: Median (Full Range); unit: days
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 6
days | 91.5 [28 to 161]

6. Secondary Outcome: Safety and Tolerability of Regimen as Measured by the Rate of the Most Common Adverse Events Experienced
Description: Adverse events will be assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Up to 13 months after start of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 51
percentage of participants
  Fatigue | 88
  Febrile neutropenia | 76
  Diarrhea | 75
  Nausea | 69

7. Secondary Outcome: Remission Duration
Description: Defined as the first date that all criteria for CR, CRi or HI are fulfilled to the date of treatment failure, relapse from CR, or death due to any cause.
Time Frame: Completion of follow-up (median follow-up was 58 months)
Population: Number of participants analyzed include those participants who met the criteria for CR, CRi, or HI.
Measure: Median (Full Range); unit: days
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 7
days | 361 [172 to 490]

8. Secondary Outcome: Progression-free Survival
Time Frame: Completion of follow-up (median follow-up was 58 months)
Population: Data was not collected for this outcome measure. Progression is very hard to define for MDS and AML and including it as a pre-specified secondary outcome measure in the protocol was an oversight.
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 0

9. Secondary Outcome: Event-free Survival
Description: Event-free survival is defined as the interval from the date of first dose of study drug to date of treatment failure, relapse from CR, or death due to any cause.
Time Frame: Completion of follow-up (median follow-up was 58 months)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 51
days | 104 [91.3 to 118]

10. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the date of first dose of study drug to the date of death from any cause.
Time Frame: Completion of follow-up (median follow-up was 58 months)
Measure: Median (Full Range); unit: months
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 51
months | 6.44 [0.2 to 63.33]

11. Secondary Outcome: Rates of Morphologic Complete Remission With Incomplete Count Recovery (CRi)
Description: Morphologic complete remission with incomplete blood count recovery (CRi): Achievement of all of the criteria for CR except for residual neutropenia (< 1,000/μL) or thrombocytopenia (< 100,000/μL).
Time Frame: Up to 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 51
percentage of participants | 3.9

12. Secondary Outcome: Rate of Hematologic Improvement.
Description: -Hematologic improvement (HI). Includes the following categories:
  * Erythroid response: Hemoglobin increase by ≥ 1.5 g/dL over baseline in which the pretreatment hemoglobin is < 11 g/dL or reduction of RBC transfusions of at least 4 RBC transfusions / 8 wk compared with the pretreatment transfusion number in the previous 8 weeks.
  * Platelet response. Absolute increase of > 30 x 10^9/L for patients starting with 20 x 10^9/L or increase from < 20 x 10^9/L to > 20 x 109/L and by at least 100%
  * Neutrophil response. At least 100% increase and an absolute increase > 0.5 x 109/L for patients with pretreatment neutrophils < 1.0 x 109/L)
Time Frame: Up to 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Level 1-Phase II (All Patients Enrolled)
Number analyzed (Participants) | 51
percentage of participants | 2.0

ADVERSE EVENTS:
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4 | Level 5 | Level 5B | Phase II
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/6 | 0/8 | 0/10 | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 6/6 | 8/8 | 10/10 | 6/6 | 14/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1 (N=4) | Level 2 (N=3) | Level 3 (N=6) | Level 4 (N=8) | Level 5 (N=10) | Level 5B (N=6) | Phase II (N=14)
ALT (Investigations) | 2 | 2 | 1 | 1 | 1 | 2 | 2
AST (Investigations) | 0 | 1 | 0 | 1 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation - mental status change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alkaline phosphatase - high (Investigations) | 0 | 0 | 0 | 3 | 1 | 0 | 4
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Allergic reaction to transfusion (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Altered mental status (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Angioedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 5 | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Arthritic hand pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus sinusitis infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atypical fungal lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Bilateral hand pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bilateral lower extremity edema (General disorders) | 0 | 0 | 0 | 4 | 5 | 0 | 0
Biopsy site pain (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 3
C. albacans infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
C. neg staph & E. faecalis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
C. neg staph & L. buccalis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 2 | 2 | 0 | 0 | 1
Chest pain (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1
Citrobacteremia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 1
Coag neg staphylococcus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coag. negative staph infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coagulase negative staphlococcus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 2 | 0 | 0 | 0 | 3 | 0 | 1
Conjunctival hemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 | 5 | 2 | 4
Creatinine (Investigations) | 2 | 2 | 0 | 2 | 4 | 1 | 2
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death due to fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 7 | 5 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Dry lips (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 2 | 2 | 5
E. Coli infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
E. Coli sepsis infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
E. Coli urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
EBV meningitis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eccymosis, right arm (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecthyma (groin) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Edema (General disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1
Edema: limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterobacter cloacae infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal line infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Enterococcus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epigastric distress (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 4
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye itch (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial edema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 2 | 2 | 2 | 6 | 6 | 6 | 7
Febrile neutropenia (Infections and infestations) | 2 | 1 | 1 | 5 | 7 | 3 | 4
Fever (General disorders) | 1 | 1 | 2 | 0 | 2 | 1 | 6
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal bacteremia/cladosporium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal pneumonia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Fungal upper respiratory infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0
GI bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2
GI upset (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 3 | 4 | 3
Generalized pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Global hypokinesis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gram negative sepsis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gram positive cocci infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HSV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 4
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 2
Hemoglobin (Blood and lymphatic system disorders) | 3 | 3 | 3 | 3 | 1 | 4 | 7
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinemia (Investigations) | 2 | 1 | 2 | 0 | 2 | 0 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 2 | 1 | 2 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 4 | 5 | 3 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 3 | 0 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1 | 6 | 1 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 1 | 4 | 3 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
INR (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 1
Ileal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incisional pain (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaw swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left hip fracture pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Left lower leg joint pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytes (Investigations) | 3 | 2 | 2 | 6 | 4 | 0 | 9
Lightheadedness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Lymphopenia (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth sores (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucositis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2 | 2 | 3
Multifocal pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (chest) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail changes; dystrophic nails (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 6 | 4 | 6
Neuropathy - fingers (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy - right chest (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy - right foot drop (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophils (Investigations) | 1 | 1 | 3 | 5 | 3 | 2 | 5
Night sweats (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Opportunistic infection NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes simplex virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral thrush infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 1
PTT (Investigations) | 2 | 0 | 0 | 1 | 2 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parainfluenza infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penis erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penumonitis, C. glabrata (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral edema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perirectal left buttock abscess/ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelets (Investigations) | 4 | 2 | 3 | 2 | 4 | 6 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Prolonged QTc interval (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prolonged intubation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pseudomonas bacteremia infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychosis - visual hallucinations (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary aspergillosis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash, actinoform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash, erythema diffuse (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Rash, macropapular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Rash, petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Restless leg syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Right lower quadrant abdomen ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rigors/chills (General disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 4
S. viridians and g+ cocci infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Saccular aneurism (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sclera discoloration blue (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Secretions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 1 | 4
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrthymia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sore/lesion on buttocks (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Splenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Submandibular gland infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Substernal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraglottal edema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supratentorial ventriculomegaly (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swollen, irritated eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 4 | 0 | 0 | 1 | 1 | 0 | 2
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Taste alteration (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tingling left leg (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheostomy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary hesitancy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urination difficult (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 1 | 5 | 2 | 4
Vulvar lesions (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Yeast infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes